CLINICAL TRIAL: NCT03027934
Title: A Single Center, Randomized, Open Label, Crossover Study With Ticagrelor and Prasugrel to Evaluate Ticagrelor Mechanism of Action in Inhibiting Juvenile Platelet ADP Response
Brief Title: A Single Center Study to Evaluate Ticagrelor Mechanism of Action in Inhibiting Juvenile Platelet ADP Response
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study population difficult to recruit
Sponsor: CirQuest Labs, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ESR-14-10619
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Drug: Ticagrelor; Drug: Prasugrel
- Group 2 (Active Comparator)
  Interventions: Drug: Ticagrelor; Drug: Prasugrel

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor, 90mg twice daily
  Other Names: Brilinta
Drug: Prasugrel — Prasurgrel, 10mg once daily
  Other Names: Effient

SUMMARY:
The overall objective of this study is to assess P2Y12 inhibition ex vivo in blood samples obtained from diabetic subjects who will be administered one of the two P2Y12 antagonists in a cross-over design.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Male or female aged 18 to 70 years, inclusive.
3. Documented current medical history of diabetes controlled by either medication or diet and/or exercise.
4. Women must have a negative urine pregnancy test.

Exclusion Criteria:

1. Pregnant or lactating females, or females of child-bearing potential (i.e., those who are not chemically or surgically sterilized or who are not post-menopause) or those who are not willing to use a medically accepted method of contraception that is considered reliable in the judgement of the investigator throughout the duration of the study or females who have a positive pregnancy test at screening.
2. Weight of less than 135 lbs.
3. Currently prescribed and taking clopidogrel (generic or Plavix), ticagrelor (Brilinta) or prasugrel (Effient) or have taken within the past 10 days.
4. Current medications:

   1. PAR-1 antagonist (vorapaxar/Zontivity) or within the last month.
   2. Phosphodiesterase inhibitors such as cilostazol (Pletal).
   3. Glycoprotein IIb/IIIa inhibitors or within the last ten days (Integrilin, Aggrastat, ReoPro).
   4. Adenosine reuptake inhibitors such as dipyridamole (Aggrenox, Persantine)
   5. Coumadin.
   6. Heparin including low molecular weight heparin.
   7. Factor Xa inhibitors (e.g., enoxaparin, rivaroxaban, apixaban, and edoxaban).
   8. Direct thrombin inhibitors (e.g., hirudin, bivalirudin, dabigatran.
   9. Concomitant therapy with strong CYP3A inhibitors, such as atanazavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazadone, nelfinavir, ritonavir, saquinavir, telithromycin, and voriconizole,
   10. Concomitant therapy with potent CYP3A inducers, such as rifampin, phenytoin, carbamazepine, and phenobarbital.
5. Increased bleeding risk including:

   1. Recent (within 30 days) GI bleeding
   2. Active pathological bleeding
   3. Any history of intracranial, intraocular, retroperitoneal, or spinal bleeding
   4. Prior history of transient ischemic attack or stroke
   5. Recent (within 3 months) major trauma
   6. Sustained uncontrolled hypertension (systolic blood pressure [SBP] > 180mmHg or diastolic blood pressure [DBP] > 100mmHg
   7. History of hemorrhagic disorders that can increase the risk of bleeding (e.g., hemophilia, von Willebrand's disease)
   8. Patients that have used within 30 days of screening, any oral or parenteral anti-thrombotic agent.
   9. Platelet count less than 100,000 mm3 or hemoglobin < 10g/dL
6. Contraindication or other reason that ticagrelor or prasugrel should not be administered (e.g., known hypersensitivity to medication or any medication component)
7. A history of alcohol and/or substance abuse that could interfere with conduct of the trial.
8. Known active or recurrent hepatic disorder (including cirrhosis, hepatitis B and hepatitis C, or confirmed (ALT/AST) levels > 3 times ULN or total bilirubin > 2 times ULN at screening.
9. Scheduled for revascularization (e.g., PCI, CABG) during the study period.
10. Any Acute Coronary Syndrome (ACS) event within the past 6 months.
11. Participation in another investigational drug or device study within 30 days of dosing.
12. Any acute or chronic unstable condition in the past 30 days or other condition which, in the opinion of the investigator, may either put the subject at risk or influence the result of the study (e.g., active cancer, risk for non-compliance, risk for lost to follow-up).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-28 (Estimated); Primary Completion 2017-10-31 (Estimated); Study Completion 2017-10-31 (Estimated)

PRIMARY OUTCOMES:
Aggregation Response | 23 hr Day 5
  Comparison of aggregation response using ADP in subjects receiving prasurgrel versus ticagrelor

SECONDARY OUTCOMES:
Reticulated Platelet Reactivity Index (PRI) | 23 hr Day 5
  Comparison of PRI as measured by VASP in subjects receiving ticagrelor versus subjects receiving prasugrel

CONTACTS AND LOCATIONS:
Overall Officials: Jayaprakash Kotha, Principal Investigator — CirQuest Labs

IPD SHARING:
Plan to Share IPD: No